CLINICAL TRIAL: NCT00630071
Title: A Prospective Study Investigating the Diagnostic Value of Procalcitonin in Patients With Acute Appendicitis
Brief Title: Diagnostic Value of Procalcitonin in Patients With Acute Appendicitis
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Dr., Ruhr University of Bochum
Other Study IDs: PCT 01
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Appendicitis
Keywords: Diagnostic Appendicitis; Procalcitonin
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1.5 ml whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The values of laboratory examinations which are useful for the diagnoses of acute appendicitis are white blood cell count (WBC), C-reactive protein (CRP) and erythrocyte blood sedimentation rate (ESR). Another laboratory value which has recently received considerable attention for the early diagnosis of bacterial infection and sepsis is pro-calcitonin (PCT). In recent studies it has been clearly shown that PCT is one of the most important biochemical indicators which closely correlates with the severity of inflammatory host response to microbial infections. Aim of this open, prospective study is therefore to investigate if PCT has an accurate diagnostic value for the diagnosis of acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of appendicitis

Exclusion Criteria:

* Antibiotic therapy
* Infection at other body sites
* Age < 14 years
* Appendectomy in the medical history

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical Emergency Room
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2008-02; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benno Mann, PD Dr. med., Study Chair — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum; Michael Sand, Dr. med., Principal Investigator — Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum
Locations (1):
- Department of General and Visceral Surgery, Augusta Krankenanstalt, Academic Teaching Hospital of the Ruhr-University Bochum, Germany, Bochum, Germany

REFERENCES:
- [Result] Sand M, Trullen XV, Bechara FG, Pala XF, Sand D, Landgrafe G, Mann B. A prospective bicenter study investigating the diagnostic value of procalcitonin in patients with acute appendicitis. Eur Surg Res. 2009;43(3):291-7. doi: 10.1159/000232939. Epub 2009 Aug 7. PMID 19672084